CLINICAL TRIAL: NCT04631666
Title: A Phase 1/2a Trial of the Intravenous Administration of the SARS-CoV-2-Neutralizing Monoclonal Antibody DZIF-10c in SARS-CoV-2-Infected and -Uninfected Individuals
Brief Title: SARS-CoV-2-Neutralizing Monoclonal COVID-19 Antibody DZIF-10c by Infusion
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: ZKS Köln (Other); Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Florian Klein, Investigator, University of Cologne
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: Uni-Koeln-4288
Record Dates: First submitted 2020-11-05; First posted 2020-11-17 (Actual); Results first posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2023-10

CONDITIONS: SARS-CoV-2 Infection
Keywords: SARS-CoV-2; Covid-19; Infusion; Monoclonal Antibody
MeSH Terms: conditions — COVID-19 | interventions — BI 767551

STUDY DESIGN:
Intervention Model Description: This study consists of an open-label dose escalation phase in healthy volunteers (Groups 1A-1C) and an additional open-label lead-in phase in SARS-CoV-2-infected individuals (Group 2C).
  After completion of the dose escalation phase, SARS-CoV-2-infected individuals will be enrolled into a randomized placebo-controlled expansion cohort (Group 2D).
  An additional higher dose cohort may be included for healthy volunteers (Group 1D).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1A (uninfected) - 2.5 mg/kg (Experimental): SARS-CoV-2-uninfected volunteers will receive a single intravenous infusion of DZIF-10c at a dose of 2.5 mg/kg
  Interventions: Biological: DZIF-10c
- Group 1B (uninfected) - 10 mg/kg (Experimental): SARS-CoV-2-uninfected volunteers will receive a single intravenous infusion of DZIF-10c at a dose of 10 mg/kg
  Interventions: Biological: DZIF-10c
- Group 1C (uninfected) - 40 mg/kg (Experimental): SARS-CoV-2-uninfected volunteers will receive a single intravenous infusion of DZIF-10c at a dose of 40 mg/kg
  Interventions: Biological: DZIF-10c
- Group 1D (uninfected) - high dose (Experimental): SARS-CoV-2-uninfected volunteers will receive a single intravenous infusion of DZIF-10c at a dose higher than 40 mg/kg
  Interventions: Biological: DZIF-10c
- Group 2C (infected) - 40 mg/kg (Experimental): SARS-CoV-2-infected volunteers will receive a single intravenous infusion of DZIF-10c at a dose of 40 mg/kg
  Interventions: Biological: DZIF-10c
- Group 2D (infected) - 40 mg/kg (Experimental): SARS-CoV-2-infected volunteers will be randomized 2:1 to receive an intravenous infusion of DZIF-10c at a dose of 40 mg/kg or placebo
  Interventions: Biological: DZIF-10c; Other: Placebo

INTERVENTIONS:
Biological: DZIF-10c — SARS-CoV-2-neutralizing monoclonal antibody DZIF-10c by intravenous infusion
Other: Placebo — Intravenous infusion of sterile normal saline (NaCl 0.9%) as placebo
  Arms: Group 2D (infected) - 40 mg/kg

SUMMARY:
This is the first-in-human phase 1/2a trial of the intravenous administration of the SARS-CoV-2-neutralizing monoclonal antibody DZIF-10c in healthy volunteers and SARS-CoV-2-infected individuals. It will evaluate the safety, pharmacokinetic profile, immunogenicity, and antiviral activity of DZIF-10c.

DETAILED DESCRIPTION:
The phase 1 component of this trial consists of a single intravenous infusion open-label dose-escalation phase (Groups 1A-1D and Group 2C). Subsequently, the highest tested and tolerated dose will be administered to an expansion cohort of SARS-CoV-2-infected individuals (Group 2D). In this randomized and blinded group, participants will receive DZIF-10c or placebo by intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

Groups 1A-1D

* Age 18-65.
* SARS-CoV-2-RNA negative naso- or oropharyngeal swab obtained within 3 calendar days before study drug administration by NAAT (e.g., qRT-PCR).
* Non-reactivity of serum antibodies (IgG; and IgA and/or IgM when tested) against SARS-CoV-2 by serological assay at screening.

Groups 2C-2D

* Age 18-70.
* SARS-CoV-2-RNA positive naso- or oropharyngeal swab obtained within 3 calendar days before study drug administration by NAAT (e.g., qRT-PCR).
* Onset of COVID-19 symptoms (e.g., sore throat, cough, fever, chills, fatigue, dys- or anosmia, dys- or ageusia, headache, muscle pain, gastrointestinal symptoms) within 7 days prior to study drug administration or Non-reactivity of serum or plasma antibodies (IgG; and IgA and/or IgM when tested) against SARS-CoV-2 by serological assay at screening.
* Disease severity score 1-4 as defined by the WHO Clinical Progression Scale (WHO, Lancet Inf Dis 2020).

Exclusion Criteria (all groups):

* Known hypersensitivity to any constituent of the investigational medicinal product.
* Hepatitis B infection indicated by detectable HBsAg (Hepatitis B surface antigen) in blood.
* Detectable antibodies against hepatitis C virus in blood unless active hepatitis C is ruled out by negative HCV-RNA.
* HIV infection indicated by detectable HIV antigen and/or HIV antibodies in blood.
* Neutrophil count ≤1,000 cells/µl
* Hemoglobin ≤10 g/dl
* Platelet count ≤100,000 cells/µl
* ALT ≥2.0 x ULN
* AST ≥2.0 x ULN
* Total bilirubin ≥1.5 ULN
* eGFR <60 ml/min/1.73m2
* Pregnancy or lactation.
* Any vaccination within 14 days prior to DZIF-10c administration.
* Receipt of any SARS-CoV-2 vaccine or SARS-CoV-2 monoclonal antibody in the past.
* Diagnosis of bronchial asthma or history of bronchial hyperresponsiveness, COPD, pulmonary fibrosis, or other chronic lung diseases.
* Any chronic or clinically significant medical condition that in the opinion of investigator would jeopardize the safety or rights of the volunteer.
* History of systemic corticosteroids, immunosuppressive anti-cancer, or other medications considered significant by the trial physician within the last 6 months (a single administration of systemic corticosteroids within ≤6 months and ≥4 weeks of enrollment is acceptable).
* Participation in another clinical trial of an investigational medicinal product within the past 12 weeks or expected participation during this study.
* Dependency on the principal investigator or study staff; or site personnel directly affiliated with this trial.
* Legally incapacitated individuals
* Individuals held in an institution by legal or official order
* If engaging in sexual activity that could result in pregnancy, inability or unwillingness to comply with the requirements for highly effective contraception

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Fätkenheuer, MD, Principal Investigator — University of Cologne
Locations (1):
- University Hospital Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kreer C, Zehner M, Weber T, Ercanoglu MS, Gieselmann L, Rohde C, Halwe S, Korenkov M, Schommers P, Vanshylla K, Di Cristanziano V, Janicki H, Brinker R, Ashurov A, Krahling V, Kupke A, Cohen-Dvashi H, Koch M, Eckert JM, Lederer S, Pfeifer N, Wolf T, Vehreschild MJGT, Wendtner C, Diskin R, Gruell H, Becker S, Klein F. Longitudinal Isolation of Potent Near-Germline SARS-CoV-2-Neutralizing Antibodies from COVID-19 Patients. Cell. 2020 Sep 17;182(6):1663-1673. doi: 10.1016/j.cell.2020.08.046. No abstract available. PMID 32946786
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Groups:
- 1A: Healthy, 2.5 mg/kg; 1B: Healthy, 10 mg/kg; 1C: Healthy, 40 mg/kg; 1D: Healthy, 80 mg/kg: Open label, SARS-CoV-2 negative, DZIF-10c i.v. infusion
- 2C: Infected, 40 mg/kg: Open label, SARS-CoV-2-infected, DZIF-10c i.v. infusion
- 2D: Infected, 40 mg/kg: Double-blind and randomized, SARS-CoV-2-infected, DZIF-10c i.v. infusion
- 2D: Infected, Placebo: Double-blind and randomized, SARS-CoV-2-infected, placebo i.v. infusion
Period: Overall Study
Arm/Group | 1A: Healthy, 2.5 mg/kg | 1B: Healthy, 10 mg/kg | 1C: Healthy, 40 mg/kg | 1D: Healthy, 80 mg/kg | 2C: Infected, 40 mg/kg | 2D: Infected, 40 mg/kg | 2D: Infected, Placebo
Started | 3 | 3 | 3 | 6 | 3 | 26 | 13
Completed | 3 | 3 | 3 | 6 | 3 | 26 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1A: Healthy, 2.5 mg/kg | 1B: Healthy, 10 mg/kg | 1C: Healthy, 40 mg/kg | 1D: Healthy, 80 mg/kg | 2C: Infected, 40 mg/kg | 2D: Infected, 40 mg/kg | 2D: Infected, Placebo | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 26 | 13 | 57
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [22 to 34] | 28 [27 to 39] | 28 [28 to 28] | 26.5 [26 to 28] | 43 [41 to 48] | 40 [30 to 52] | 32 [25 to 47] | 32 [27.5 to 42.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 1 | 5 | 2 | 11 | 5 | 27
  Male | 3 | 0 | 2 | 1 | 1 | 15 | 8 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 3 | 3 | 3 | 6 | 3 | 26 | 13 | 57

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Any AE Within 7 d of Study Drug Infusion
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Healthy, 2.5 mg/kg | 1B: Healthy, 10 mg/kg | 1C: Healthy, 40 mg/kg | 1D: Healthy, 80 mg/kg | 2C: Infected, 40 mg/kg | 2D: Infected, 40 mg/kg | 2D: Infected, Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 26 | 13
Participants | 2 | 1 | 0 | 0 | 0 | 11 | 8

2. Secondary Outcome: DZIF-10c Elimination Half Life
Description: DZIF-10c serum elimination half-life
Time Frame: 0, 1, and 4 hours post dose; 1, 3, 7, 14, 21, 28, 56, 90 days post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | 1A: Healthy, 2.5 mg/kg | 1B: Healthy, 10 mg/kg | 1C: Healthy, 40 mg/kg | 1D: Healthy, 80 mg/kg | 2C: Infected, 40 mg/kg | 2D: Infected, 40 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 26
days | 28.4 (17.5) | 24.2 (12.8) | 20.1 (9.53) | 20.9 (25.4) | 16.8 (45) | 21.8 (12.2)

3. Secondary Outcome: DZIF-10c Peak Serum Concentration
Time Frame: 0, 1, and 4 hours post dose; 1, 3, 7, 14, 21, 28, 56, 90 days post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/ml
Arm/Group | 1A: Healthy, 2.5 mg/kg | 1B: Healthy, 10 mg/kg | 1C: Healthy, 40 mg/kg | 1D: Healthy, 80 mg/kg | 2C: Infected, 40 mg/kg | 2D: Infected, 40 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 26
µg/ml | 54.3 (12.6) | 207 (8.92) | 738 (7.94) | 1480 (10.2) | 983 (8.9) | 970 (21.5)

4. Secondary Outcome: DZIF-10c Area Under the Curve
Description: Area under the curve based on serum antibody levels
Time Frame: 0, 1, and 4 hours post dose; 1, 3, 7, 14, 21, 28, 56, 90 days post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg h/ml
Arm/Group | 1A: Healthy, 2.5 mg/kg | 1B: Healthy, 10 mg/kg | 1C: Healthy, 40 mg/kg | 1D: Healthy, 80 mg/kg | 2C: Infected, 40 mg/kg | 2D: Infected, 40 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 26
µg h/ml | 15400 (5.79) | 61700 (14.3) | 212000 (18.9) | 358000 (14) | 236000 (24.4) | 235000 (15.5)

5. Secondary Outcome: DZIF-10c Clearance
Time Frame: 0, 1, and 4 hours post dose; 1, 3, 7, 14, 21, 28, 56, 90 days post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ml/day
Arm/Group | 1A: Healthy, 2.5 mg/kg | 1B: Healthy, 10 mg/kg | 1C: Healthy, 40 mg/kg | 1D: Healthy, 80 mg/kg | 2C: Infected, 40 mg/kg | 2D: Infected, 40 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 23
ml/day | 311 (10.6) | 242 (26.8) | 282 (40.8) | 341 (14.1) | 280 (24.2) | 339 (20.6)

6. Secondary Outcome: DZIF-10c Volume of Distribution Vz
Time Frame: 0, 1, and 4 hours post dose; 1, 3, 7, 14, 21, 28, 56, 90 days post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ml
Arm/Group | 1A: Healthy, 2.5 mg/kg | 1B: Healthy, 10 mg/kg | 1C: Healthy, 40 mg/kg | 1D: Healthy, 80 mg/kg | 2C: Infected, 40 mg/kg | 2D: Infected, 40 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 26
ml | 12800 (11.7) | 8460 (18) | 8160 (45.7) | 10300 (21.8) | 6790 (29.6) | 10700 (19.7)

7. Secondary Outcome: Anti-Drug Antibody Development
Description: Individuals developing anti-drug antibodies
Time Frame: 0, 14, 28, 56, 90 days post dose
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Healthy, 2.5 mg/kg | 1B: Healthy, 10 mg/kg | 1C: Healthy, 40 mg/kg | 1D: Healthy, 80 mg/kg | 2C: Infected, 40 mg/kg | 2D: Infected, 40 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 26
Participants | 0 | 0 | 0 | 0 | 1 | 0

8. Secondary Outcome: Anti-Drug Antibody Peak Titer
Description: Magnitude of the development of anti-drug antibodies targeting DZIF-10c in individuals developing such antibodies (peak serum titer)
Time Frame: 0, 14, 28, 56, 90 days post dose
Measure: Number; unit: reciprocal serum titer
Arm/Group | 2C: Infected, 40 mg/kg
Number analyzed (Participants) | 1
reciprocal serum titer | 960

9. Secondary Outcome: Time-weighted SARS-CoV-2 Viral Load Change From Baseline
Description: Time-weighted change of SARS-CoV-2 viral load from baseline in nasopharyngeal swab samples as determined by the SARS-CoV-2 E gene; based on a parametric analysis of covariance model with corresponding baseline viral load, antibody status at baseline, and treatment; determined as the adjusted mean area over the curve (AOC) for samples collected at baseline and 1, 3, 7, 14, 28 days post dose
Time Frame: 0, 1, 3, 7, 14, 28 days post dose
Measure: Mean (Standard Error); unit: log10 cp/ml
Arm/Group | 2D: Infected, 40 mg/kg | 2D: Infected, Placebo
Number analyzed (Participants) | 26 | 13
log10 cp/ml
  Over 7 days | -2.035 (0.146) | -1.449 (0.217)
  Over 14 days | -3.273 (0.126) | -2.668 (0.188)
  Over 28 days | -3.938 (0.096) | -3.576 (0.143)

10. Secondary Outcome: MMRM SARS-CoV-2 Viral Load Change From Baseline
Description: Change of SARS-CoV-2 viral load from baseline in nasopharyngeal swab samples as determined by the SARS-CoV-2 E gene; based on Mixed Model for Repeated Measures (MMRM) with fixed effects for antibody status at BL, LOG10 (viral load) at BL and interaction with visit, treatment-by-visit interaction, and random effect for patient; samples collected at baseline and 1, 3, 7, 14, 28 days post dose
Time Frame: 0, 1, 3, 7, 14, 28 days post dose
Measure: Mean (Standard Error); unit: Adjusted log10 cp/ml
Arm/Group | 2D: Infected, 40 mg/kg | 2D: Infected, Placebo
Number analyzed (Participants) | 26 | 13
Adjusted log10 cp/ml
  Over 7 days | -4.3 (0.2) | -3.3 (0.3)
  Over 14 days | -4.5 (0.2) | -4.3 (0.3)
  Over 28 days | -4.7 (0.1) | -4.6 (0.1)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events: All adverse events after drug intake until final study visit (Day 90 visit)
Description: Participants were queried for Adverse Events at all study visits
Groups:
- 1A: Healthy, 2.5 mg/kg: SARS-CoV-2-uninfected volunteers will receive a single intravenous infusion of DZIF-10c at a dose of 2.5 mg/kg
  DZIF-10c: SARS-CoV-2-neutralizing monoclonal antibody DZIF-10c by intravenous infusion
- 1B: Healthy, 10 mg/kg: SARS-CoV-2-uninfected volunteers will receive a single intravenous infusion of DZIF-10c at a dose of 10 mg/kg
  DZIF-10c: SARS-CoV-2-neutralizing monoclonal antibody DZIF-10c by intravenous infusion
- 1C: Healthy, 40 mg/kg: SARS-CoV-2-uninfected volunteers will receive a single intravenous infusion of DZIF-10c at a dose of 40 mg/kg
  DZIF-10c: SARS-CoV-2-neutralizing monoclonal antibody DZIF-10c by intravenous infusion
- 1D: Healthy, 80 mg/kg: SARS-CoV-2-uninfected volunteers will receive a single intravenous infusion of DZIF-10c at a dose higher than 40 mg/kg
  DZIF-10c: SARS-CoV-2-neutralizing monoclonal antibody DZIF-10c by intravenous infusion
- 2C: Infected, 40 mg/kg: SARS-CoV-2-infected volunteers will receive a single intravenous infusion of DZIF-10c at a dose of 40 mg/kg
  DZIF-10c: SARS-CoV-2-neutralizing monoclonal antibody DZIF-10c by intravenous infusion
- 2D: Infected, 40 mg/kg: SARS-CoV-2-infected volunteers randomized to receive an intravenous infusion of DZIF-10c at a dose of 40 mg/kg (blinded)
  DZIF-10c: SARS-CoV-2-neutralizing monoclonal antibody DZIF-10c by intravenous infusion
- 2D: Infected, Placebo: SARS-CoV-2-infected volunteers randomized to receive an intravenous infusion of placebo (blinded)
  Placebo: Sterile normal saline
Arm/Group | 1A: Healthy, 2.5 mg/kg | 1B: Healthy, 10 mg/kg | 1C: Healthy, 40 mg/kg | 1D: Healthy, 80 mg/kg | 2C: Infected, 40 mg/kg | 2D: Infected, 40 mg/kg | 2D: Infected, Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/6 | 0/3 | 0/26 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/6 | 0/3 | 0/26 | 0/13
Other Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 2/3 | 0/6 | 1/3 | 18/26 | 10/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1A: Healthy, 2.5 mg/kg (N=3) | 1B: Healthy, 10 mg/kg (N=3) | 1C: Healthy, 40 mg/kg (N=3) | 1D: Healthy, 80 mg/kg (N=6) | 2C: Infected, 40 mg/kg (N=3) | 2D: Infected, 40 mg/kg (N=26) | 2D: Infected, Placebo (N=13)
Flushing (Vascular disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0 | 0 | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 8 (10) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 (4) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Headache (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 8 (9) | 5 (5)
Hyposmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 2 (2)
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2)
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 4 (4) | 2 (2)
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1)
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 | 0 | 0 | 0 | 1 (1) | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
COVID-19 (Infections and infestations) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications by PIs are to be submitted to the sponsor for review at least 30 days prior to planned disclosure. Modifications suggested by the sponsor should be considered unless they affect the scientific character or neutrality of the publication. A maximum embargo period of 90 days is applicable only if disclosure would affect (potential) intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT04631666/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT04631666/SAP_001.pdf